CLINICAL TRIAL: NCT07011953
Title: A Clinical Trial of Adjunctive Thyroxine for Avolition in Schizophrenia
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xin Yu, Professor, Peking University
Allocation: Not Applicable | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-06-02
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Schizophrenia; Avolition
Keywords: schizophrenia; avolition; thyroxine; double blind; randomized controlled trial; motivation
MeSH Terms: conditions — Schizophrenia | interventions — Antipsychotic Agents; Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group: adjunctive thyroxine (Experimental): Maintain the original antipsychotic regimen combined with levothyroxine sodium tablets (Euthyrox), 50 μg/day for 8 weeks. Manufacturer: Merck Serono Ltd.
  Interventions: Drug: Antipsychotics plus Levothyroxine Sodium
- Placebo Control group (Placebo Comparator): The placebo control group will maintain the original antipsychotic regimen, supplemented with a dose-equivalent placebo tablet (starch tablet) matching levothyroxine sodium in appearance and nominal dosage (50 μg/day) for 8 weeks. Manufacturer: Boji Medical Technology Co., Ltd.
  Interventions: Drug: Antipsychotics plus Placebo

INTERVENTIONS:
Drug: Antipsychotics plus Levothyroxine Sodium — Maintain the original antipsychotic regimen combined with levothyroxine sodium tablets (Euthyrox), 50 μg/day for 8 weeks. Manufacturer: Merck Serono Ltd. Levothyroxine Sodium Tablets should be administered as a single daily dose on an empty stomach, 30 minutes before breakfast, with sufficient liquid (e.g., half a glass of water).
  Arms: Treatment group: adjunctive thyroxine
Drug: Antipsychotics plus Placebo — All participants maintain pre-study antipsychotic medication at stable doses. ADDITIONALLY, they receive a visually identical placebo tablet.
  Placebo characteristics & Blinding guaranteet: Matches levothyroxine in appearance (size/color/coating), taste, and packaging.
  Active ingredien : starch tablet with no biological activity. Administration: Once daily in the morning under identical fasting conditions.
  Arms: Placebo Control group

SUMMARY:
The goal of this clinical trial is to investigate whether adjunctive thyroxine treatment can ameliorate motivation deficits in adults with schizophrenia experiencing predominant avolition (core negative symptom).

The main questions it aims to answer are:

* Does adjunctive thyroxine reduce avolition symptoms compared to placebo?
* Does adjunctive thyroxine normalize cortico-striatal circuit activity during reward processing?

Researchers will compare the treatment group (adjunctive sodium tablets, 50μg/day) with the control group (dose-equivalent placebo starch tablet) to see if thyroid hormone:

1. Significantly improves clinical scores of avolition
2. Modulates neural activation in motivation-processing brain circuits

Participants will:

* Maintain stable antipsychotic therapy for 8 weeks
* Receive daily levothyroxine/placebo tablets
* Complete the following assessments pre-/post-treatment:
* Clinical evaluations (PANSS, NSA, PSP)
* MRI scans (resting-state, structural, fMRI during reward tasks)
* Blood tests
* Behavioral motivation tasks

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for schizophrenia according to the International Classification of Diseases, 10th Revision (ICD-10) (World Health Organization, 1993);
2. Aged between 18 and 45 years, right-handed;
3. Currently clinically stable, with the primary antipsychotic medication formulation and dosage unchanged for at least 4 weeks, and a total PANSS score ≤ 60;
4. Predominant avolition symptoms, defined as a score ≥ 16 on the Motivation subscale of the Negative Symptom Assessment (NSA-15) (Zhou et al., 2023), with fewer than 3 items scoring ≥ 4 and fewer than 2 items scoring ≥ 5 on the PANSS positive subscale (Rabinowitz et al., 2013);
5. Receiving one or two second-generation antipsychotics (SGAs), with stable medication doses for at least 1 month;
6. Willingness and ability to maintain stable medication doses throughout the trial period;
7. Capacity to understand study procedures, cooperate with all testing requirements, and provide written informed consent.

Exclusion Criteria:

1. Current treatment with clozapine or first-generation antipsychotics;
2. Current use of thyroid hormone medications or presence of thyroid dysfunction;
3. Hypersensitivity to levothyroxine sodium; or history of non-hypothyroid-related heart failure, tachyarrhythmias, or recent myocardial infarction;
4. Current use of medications known to interact with levothyroxine sodium that may affect its efficacy or safety (e.g., antidiabetic drugs, coumarin derivatives);
5. History of endocrinological or cardiovascular/cerebrovascular diseases;
6. IQ < 80 assessed by the Chinese short-form Wechsler Adult Intelligence Scale (Gong, 1981);
7. History of substance abuse or drug addiction;
8. History of traumatic brain injury or neurological disorders;
9. Receiving electroconvulsive therapy (ECT) within the last 3 months;
10. Pregnancy, lactation, or planning pregnancy within the next 2 months (for female participants);
11. Claustrophobia; implanted metal devices (e.g., prosthetic implants, pacemakers); or other contraindications to MRI scanning.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
the score of Motivation subscale of the Negative Symptom Assessment (NSA-15) | Baseline, 2-week follow-up, 4-week follow-up, 6-week follow-up, 8-week follow-up

SECONDARY OUTCOMES:
Motivational deficits(avolition) measured by N2 (Emotional Withdrawal) and N4 (Passive/Apathetic, Social Withdrawal) items in the Positive and Negative Syndrome Scale (PANSS). | Baseline, 2-week follow-up, 4-week follow-up, 6-week follow-up, 8-week follow-up
Performance of the monetary incentive delay task (MID) | baseline, 8-week follow-up
Performance of the Effort-Expenditure for Rewards Task (EEfRT) | baseline, 8-week follow-up